#### The GlaxoSmithKline group of companies

| Division | : | Worldwide Development |
|------------------|---|-----------------------------------|
| Information Type | : | Reporting and Analysis Plan (RAP) |

| Title | ÷ | Reporting and Analysis Plan for Study 205893: A 2-Part Phase I, Single Dose, Crossover Relative Bioavailability Study of Both TIVICAY 10 mg Conventional Tablets and 5 mg Dispersible Tablets Compared to Conventional TIVICAY Tablets in Healthy Adult Subjects |
|---|---|---|
| <b>Compound Number</b> | : | GSK1349572 |
| <b>Effective Date</b> | : | 19-JUN-2017 |

#### **Description:**

- The purpose of this RAP is to describe the planned analyses and output to be included in the Clinical Study Report for Protocol 205893.
- This RAP is intended to describe the safety, tolerability, and pharmacokinetic (PK) analyses required for the study.
- This RAP will be provided to the study team members to convey the content of the Statistical Analysis Complete (SAC) deliverable.

#### **Author's Name and Functional Area:**

| PPD | 25-JUN-2017 |
|---|---|
| Biostatistician II (Biostatistics, Early Development Services, PPD) | 23-JUIN-201/ |
| PPD | 25 HIN 2017 |
| Pharmacokineticist (Biostatistics, PPD) | 25-JUN-2017 |

#### Approved by:

| PPD | | 25-JUN-2017 |
|-----------------|--------------------------------------------|-------------|
| Manager (Statis | stics, Programming and Data Strategy, GSK) | 23-JUN-2017 |

Copyright 2017 the GlaxoSmithKline group of companies. All rights reserved. Unauthorised copying or use of this information is prohibited.

#### **TABLE OF CONTENTS**

| | | | | PAGE |
|---|---|---|---|---|
| 1. | REPO | RTING & | ANALYSIS PLAN SYNPOSIS | 4 |
| 2. | SUMM<br>2.1.<br>2.2.<br>2.3.<br>2.4. | Changes<br>Study O<br>Study D | KEY PROTOCOL INFORMATION s to the Protocol Defined Statistical Analysis Plan bjective(s) and Endpoint(s) esign al Hypotheses | 7<br>7 |
| 3. | PLANI<br>3.1. | | ALYSESalyses | |
| 4. | ANAL` | | PULATIONS | |
| 5. | | | ONS FOR DATA ANALYSES AND DATA HANDLING S | 12 |
| 6. | STUD 6.1. | | ATION ANALYSESw of Planned Analyses | |
| 7. | PRIMA<br>7.1. | | TISTICAL ANALYSES | |
| 8. | SECO<br>8.1.<br>8.2. | Safety A | STATISTICAL ANALYSESanalysestory Analyses | 17 |
| 9. | REFE | RENCES | | 19 |
| 10. | 10.1. | Appendi<br>10.1.1. | | 21<br>21 |
| | 10.2. | Appendi<br>10.2.1. | ix 2: Treatment States and Phases Treatment States | 22 |
| | 10.3. | Appendi<br>10.3.1.<br>10.3.2. | ix 3: Data Display Standards & Handling Conventions Study Treatment & Sub-group Display Descriptors | 23<br>23 |

| | | 10.3.2.2. | Derivations and Handling of Missing Baseline | |
|---|---|---|---|---|
| | | | Data | 24 |
| | 10.3.3. | Reporting | Process & Standards | 24 |
| 10.4. | <b>Appendix</b> | | and Transformed Data | |
| | 10.4.1. | General | | 27 |
| | 10.4.2. | Study Pop | ulation | 27 |
| | 10.4.3. | Safety | | 27 |
| 10.5. | <b>Appendix</b> | 5: Premati | ure Withdrawals & Handling of Missing Data | 29 |
| | 10.5.1. | | Withdrawals | |
| | 10.5.2. | Handling o | f Missing Data | 29 |
| | | 10.5.2.1. | Handling of Missing Dates | 29 |
| | | 10.5.2.2. | Handling of Partial Dates | 30 |
| 10.6. | <b>Appendix</b> | 6: Values | of Potential Clinical Importance | 31 |
| | 10.6.1. | | | |
| | 10.6.2. | Vital Signs | | 31 |
| 10.7. | Appendix | 7: Multiple | Comparisons & Multiplicity | 32 |
| | 10.7.1. | Handling o | of Multiple Comparisons & Multiplicity | 32 |
| 10.8. | Appendix | | Checking and Diagnostics for Statistical | |
| | | | | 33 |
| 10.9. | | | viations & Trade Marks | |
| | | | ons | |
| | | | (S | |
| 10.10. | Appendix | 10: List of | Data Displays | 36 |
| | | | nple Shell Referencing | |
| | | | e [Priority] | |
| | 10.10.3. | Study Pop | ulation Tables | 37 |
| | 10.10.4. | | oles | |
| | 10.10.5. | • | kinetic Tables | |
| | 10.10.6. | Pharmacol | kinetic Figures | 40 |
| | | | y Tables | |
| | | | ,<br>1S | |

# 1. REPORTING & ANALYSIS PLAN SYNPOSIS

| Overview | Key Elements of the RAP |
|---|---|
| Purpose | The purpose of this reporting and analysis plan (RAP) is to describe any planned analyses and output to be included in the clinical study report for Protocol 205893. |
| Protocol | This RAP is based on the original protocol (Dated: 23/FEB/2017) of study 205893 (GSK Document No. 2016N302761_00). |
| Primary | Part 1: |
| Objective | To evaluate the relative bioavailability (BA) of dolutegravir (DTG) conventional 10 mg tablets (5 tablets) administered direct to mouth as compared to a conventional 50 mg tablet (reference) administered direct to mouth. |
| | Part 2: |
| | To evaluate the relative BA of DTG dispersible 5-mg tablets (5 tablets) administered as "disperse and immediately take" and of DTG dispersible 5-mg tablets (5 tablets) administered direct to mouth as compared to a conventional 25 mg tablet (reference) administered direct to mouth. |
| Primary | Parts 1 and 2: |
| Endpoint | Plasma DTG AUC(0-∞), AUC(0-t), and Cmax. |
| Secondary | Part 1: |
| Objectives | To compare the single dose PK of DTG conventional 10 mg tablets (5 tablets) administered direct to mouth as compared to a conventional 50 mg tablet (reference) administered direct to mouth. |
| | To evaluate the safety and tolerability of DTG conventional 10 mg (5 tablets) administered direct to mouth as compared to the administration of a conventional 50 mg tablet (reference) administered direct to mouth. |
| | Part 2: |
| | To compare the single dose PK of DTG dispersible 5-mg tablets (5 tablets) administered as "disperse and immediately take" and of DTG dispersible 5-mg tablets (5 tablets) administered direct to mouth as compared to a conventional 25 mg tablet (reference) administered direct to mouth. |
| | To evaluate the safety and tolerability of DTG dispersible 5-mg tablets (5 tablets) administered as "disperse and immediately take" and of DTG dispersible 5-mg tablets (5 tablets) administered direct to mouth as compared to a conventional 25 mg tablet (reference) administered direct to mouth. |
| Secondary | Parts 1 and 2: |
| Endpoints | <ul> <li>Plasma DTG tlag, tmax, t½, λz, %AUCex, AUC0-24, CL/F and Vz/F, Ct, and C24.</li> </ul> |
| | Safety and tolerability parameters as assessed by change from baseline in |

| Overview | Key Elements of the RAP |
|---|---|
| | number of subjects with adverse events (AEs) and Division of Acquired Immune Deficiency Syndrome (DAIDS) toxicity grading for HIV-infected patients of clinical laboratory tests. |
| Exploratory Objective | To evaluate the palatability of the dispersible tablets (Part 2 only). |
| Exploratory Endpoint | Palatability Questionnaire (Part 2 only). |
| Study<br>Design | <ul> <li>This study will be conducted as a 2-part, open-label, randomized, cross-over<br/>design with one group of subjects in Part 1 of the study randomized to receive<br/>each of 2 study treatments (A and B) over 2 dosing periods, and another group<br/>of subjects in Part 2 of the study randomized to receive each of 3 study<br/>treatments (C, D, and E) over 3 dosing periods. Treatments are defined below:</li> </ul> |
| | <ul> <li>Treatment A: Conventional 10-mg DTG tablet (5 tablets, test) administered<br/>direct to mouth.</li> </ul> |
| | <ul> <li>Treatment B: Conventional 50-mg DTG tablet (reference) administered<br/>direct to mouth.</li> </ul> |
| | <ul> <li>Treatment C: 5-mg dispersible DTG tablet (5 tablets) administered as a<br/>dispersion and immediately taken (test 1).</li> </ul> |
| | <ul> <li>Treatment D: 5-mg dispersible DTG tablet (5 tablets) administered as direct<br/>to mouth (test 2).</li> </ul> |
| | <ul> <li>Treatment E: Conventional 25-mg DTG tablet administered as direct to<br/>mouth (reference).</li> </ul> |
| | <ul> <li>Subjects will participate in only one part of the study. Parts 1 and 2 of the study may be conducted concurrently. There will be a washout of at least 7 (-4 hours) days between doses of study medication. Note: The -4 hours is an allowed tolerance window to the 7 day washout and is to allow the study site and subjects flexibility in scheduling admission and dosing for subsequent treatment periods (i.e., treatment periods 2 and/or 3).</li> </ul> |
| | <ul> <li>Part 1 is a 2-period, cross-over study that will assess the relative BA of DTG conventional 10 mg tablets (5 tablets) administered direct to mouth as compared to a conventional 50 mg tablet (reference) administered direct to mouth (treatments A and B, respectively). Each subject will receive both treatments according to their assigned treatment sequence (AB or BA)</li> </ul> |
| | <ul> <li>Part 2 is a 3-period, cross-over study that will assess the relative BA of DTG dispersible 5-mg tablets (5 tablets) administered as "disperse and immediately take" and of DTG dispersible 5-mg tablets (5 tablets) administered direct to mouth as compared to a conventional 25 mg tablet (reference) administered direct to mouth (treatments C, D, and E, respectively). Each subject will receive all three treatments according to their assigned treatment sequence (CDE, DEC, ECD, CED, DCE, or EDC).</li> </ul> |
| Planned<br>Analyses | Plasma DTG concentration-time data will be analyzed by non-compartmental methods with Phoenix WinNonlin. Calculations will be based on the actual |

| Overview | Key Elements of the RAP |
|---|---|
| | sampling times recorded during the study. From the plasma concentration-time data, the following PK parameters will be determined, as data permit: AUC(0-∞), area under the plasma concentration-time curve from time of dose to last measurable concentration (AUC(0-t)), area under the plasma concentration-time curve from time of dose to 24 hr (AUC0-24), maximum observed concentration (Cmax), plasma DTG lag time for absorption (tlag), time of occurrence of Cmax (tmax), terminal elimination phase half-life (t1/2), terminal rate constant (λz), %AUCex, apparent oral clearance (CL/F) and apparent volume of distribution during terminal phase (Vz/F), Ct, and concentration at 24 hours after dose administration (C24). |
| | Pharmacokinetic data will be listed and may be presented in graphical form and will be summarized descriptively. All PK data will be stored in the Archives, GlaxoSmithKline Research and Development (R&D) or their designee. |
| | The PK parameters except tmax and tlag) will be In-transformed and separately analyzed using a mixed effects model with fixed effect terms for period and treatment for each treatment comparison. Subject will be treated as a random effect in the model. Point estimates and their associated 90% confidence intervals (CIs) will be constructed for the differences in PK parameter values between test and reference treatments. The point estimates and their associated 90% CIs will then be back-transformed to provide point estimates and 90% CIs for the ratios of PK parameters between test and reference treatments. |
| | Safety data will be presented in tabular format and summarized descriptively according to GSK's Integrated Data Standards Library (IDSL) standards. No formal statistical analysis of the safety data will be conducted. |
| | Palatability questionnaire variables will be summarized descriptively. |
| Analysis<br>Populations | All Subjects Population: all subjects who receive at least one dose of study medication. This population will be used for all demographic and safety summaries |
| | PK Population: subjects in the 'All Subjects' population for whom a PK sample was obtained and had evaluable PK assay results. PK samples that may be affected by protocol deviations will be reviewed by the study team to determine whether or not the sample will be excluded. This population will be used for reporting of PK data. |
| Hypothesis | This study is designed to estimate the relative BA of each test treatment to the reference treatment (A vs. B; C vs. E and D vs. E) in both study parts in the fasted state. |
| | No formal hypothesis will be tested. For each pharmacokinetic endpoint (except for time of occurrence of Cmax [tmax] and tlag), point estimates and corresponding 90% Cls will be constructed for the ratio of the geometric mean of the test treatment to the geometric mean of the reference treatment, $\mu(\text{test})/\mu(\text{reference})$ . |

#### 2. SUMMARY OF KEY PROTOCOL INFORMATION

#### 2.1. Changes to the Protocol Defined Statistical Analysis Plan

The parameter "t" in the list of secondary endpoints in the protocol has been excluded as this does not represent an actual PK parameter and may be a typographical error in the protocol text. There were no other changes to or deviations from the originally planned statistical analysis specified in the protocol (Dated: 23/FEB/2017).

Listings of clinical laboratory data above a certain DAIDs toxicity grading are included in the outputs. Section 3.3.1 of the protocol indicated that these listings contain toxicities of grade 3 or higher; however, the listings will instead contain toxicities of grade 2 or higher.

#### 2.2. Study Objective(s) and Endpoint(s)

| Objectives | Endpoints |
|---|---|
| Primary Objectives | Primary Endpoints |
| Part 1 | Part 1 |
| To evaluate the relative BA of DTG conventional 10 mg tablets (5 tablets) administered direct to mouth as compared to a conventional 50 mg tablet (reference) administered direct to mouth. | Plasma DTG AUC(0-∞), AUC(0-t), and Cmax. |
| Part 2 | Part 2 |
| To evaluate the relative BA of DTG dispersible 5-mg tablets (5 tablets) administered as "disperse and immediately take" and of DTG dispersible 5-mg tablets (5 tablets) administered direct to mouth as compared to a conventional 25 mg tablet (reference) administered direct to mouth. | Plasma DTG AUC(0-∞), AUC(0-t), and Cmax. |
| Secondary Objectives | Primary Objectives |
| Part 1 | Part 1 |
| To compare the single dose PK of DTG conventional 10 mg tablets (5 tablets) administered direct to mouth as compared to a conventional 50 mg tablet (reference) administered direct to mouth. | <ul> <li>Plasma DTG tlag, tmax, t½, λz, %AUCex, AUC0-24, CL/F and Vz/F, Ct, and C24.</li> <li>Safety and tolerability parameters as assessed by change from baseline in number of subjects with AEs and DAIDS toxicity grading for HIV-infected patients of clinical laboratory tests as described in Appendix</li> </ul> |

| Objectives | Endpoints |
|---|---|
| To evaluate the safety and tolerability of DTG conventional 10 mg (5 tablets) administered direct to mouth as compared to the administration of a conventional 50 mg tablet (reference) administered direct to mouth. | 6 of the protocol. |
| <ul> <li>To compare the single dose PK of DTG dispersible 5-mg tablets (5 tablets) administered as "disperse and immediately take" and of DTG dispersible 5 mg tablets (5 tablets) administered direct to mouth as compared to a conventional 25 mg tablet (reference) administered direct to mouth.</li> <li>To evaluate the safety and tolerability of DTG dispersible 5-mg tablets (5 tablets) administered as "disperse and immediately take" and of DTG dispersible 5 mg tablets (5 tablets) administered direct to mouth as compared to a conventional 25 mg tablet (reference) administered direct to mouth.</li> </ul> | <ul> <li>Plasma DTG tlag, tmax, t½, λz, %AUCex, AUC0-24, CL/F and Vz/F, Ct, and C24.</li> <li>Safety and tolerability parameters as assessed by change from baseline in number of subjects with AEs and DAIDS toxicity grading for HIV-infected patients of clinical laboratory tests as described in Appendix 6 of the protocol.</li> </ul> |
| Exploratory Objectives | Exploratory Endpoints |
| Part 2 only | Part 2 only |
| To evaluate the palatability of the dispersible tablets. | Palatability Questionnaire. |

#### 2.3. Study Design



| Overview of S | Overview of Study Design and Key Features |
|---|---|
| | Treatment D: 5-mg dispersible DTG tablet (5 tablets) administered as direct to mouth (test 2). |
| | Treatment E: Conventional 25-mg DTG tablet administered as direct to mouth (reference). |
| Treatment | Part 1: |
| Assignment | <ul> <li>On Period 1 Day 1, subjects will be randomized to one of the 2 following<br/>treatment sequences: AB or BA in accordance with the randomization<br/>schedule generated prior to the start of the study, using validated software.</li> <li>Part 2:</li> </ul> |
| | On Period 1 Day 1, subjects will be randomized to one of the 6 following treatment sequences: CDE, DEC, ECD, CED, DCE, or EDC in accordance with the randomization schedule generated prior to the start of the study, using validated software. |
| Interim<br>Analysis | There will be no interim analysis. |

### 2.4. Statistical Hypotheses

This study is designed to estimate the relative BA of each test treatment to the reference treatment (A vs. B; C vs. E and D vs. E) in both study parts in the fasted state.

No formal hypothesis will be tested. For each pharmacokinetic endpoint (except for time of occurrence of Cmax [tmax] and tlag), point estimates and corresponding 90% CIs will be constructed for the ratio of the geometric mean of the test treatment to the geometric mean of the reference treatment,  $\mu(\text{test})/\mu(\text{reference})$ .

#### 3. PLANNED ANALYSES

#### 3.1. Final Analyses

The final planned primary analyses will be performed after the completion of the following sequential steps:

- 1. All subjects have completed the study as defined in the protocol
- 2. All required database cleaning activities have been completed and final database release and database freeze has been declared by Data Management.

#### 4. ANALYSIS POPULATIONS

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| All Subjects | <ul> <li>All subjects who receive at least one dose of<br/>study medication.</li> </ul> | <ul><li>Demographic</li><li>Safety</li></ul> |
| PK | Subjects in the "All Subjects" population for<br>whom a PK sample was obtained and had<br>evaluable PK assay results. PK samples that<br>may be affected by protocol deviations will be<br>reviewed by the study team to determine | • PK |

| Population | Definition / Criteria | Analyses Evaluated |
|---|---|---|
| | whether or not the sample will be excluded. | |

#### NOTES:

• Please refer to Appendix 10: List of Data Displays which details the population to be used for each display being generated.

#### 4.1. Protocol Deviations

- Important protocol deviations (including deviations related to study inclusion/exclusion criteria, conduct of the trial, patient management or patient assessment) will be summarised and listed.
- Protocol deviations will be tracked by the study team throughout the conduct of the study in accordance with the Protocol Deviation Management Plan.
  - Data will be reviewed prior to freezing the database to ensure all important deviations and deviations which may lead to exclusion from the analysis are captured and categorised on the protocol deviations dataset.
  - This dataset will be the basis for the summaries and listings of protocol deviations.
- A separate summary and listing of all inclusion/exclusion criteria deviations will also be provided. This summary will be based on data as recorded on the inclusion/exclusion page of the electronic case report form (eCRF).

# 5. CONSIDERATIONS FOR DATA ANALYSES AND DATA HANDLING CONVENTIONS

Table 1 provides an overview of appendices within the RAP for outlining general considerations for data analyses and data handling conventions.

Table 1 Overview of Appendices

| Section | Component |
|---|---|
| 10.1 | Appendix 1: Time & Events |
| 10.2 | Appendix 2: Treatment States and Phases |
| 10.3 | Appendix 3: Data Display Standards & Handling Conventions |
| 10.4 | Appendix 4: Derived and Transformed Data |
| 10.5 | Appendix 5: Premature Withdrawals & Handling of Missing Data |
| 10.6 | Appendix 6: Values of Potential Clinical Importance |
| 10.7 | Appendix 7: Multiple Comparisons and Multiplicity |
| 10.8 | Appendix 8: Model Checking and Diagnostics for Statistical Analyses. |
| 10.9 | Appendix 9: Abbreviations and Trade Marks |
| 10.10 | Appendix 10: List of Data Displays |

#### 6. STUDY POPULATION ANALYSES

## 6.1. Overview of Planned Analyses

The study population analyses will be based on the "All Subjects" population, unless otherwise specified.

Table 2 provides an overview of the planned study population analyses, with full details of data displays being presented in Appendix 10: List of Data Displays.

Table 2 Overview of Planned Study Population Analyses

| Display Type | Data Display | Data Display's Generated | |
|---|---|---|---|
| | Figure | Table | Listing |
| Enrollment | | | |
| Number of Subjects Enrolled by Country and Site ID | | Y | |
| Randomisation | | | |
| Randomisation | | | Υ |
| Subject Disposition | | | |
| Subject Disposition | | Υ | |
| Reasons for Screening Failures | | Υ | Υ |
| Reasons for Withdrawals | | | Υ |
| Important Protocol Deviations | | Υ | Υ |
| Inclusion and Exclusion Criteria Deviations | | | Υ |
| Demography | | | |
| Demographics Characteristics | | Y | Υ |
| Race and Racial Combinations | | Y | Υ |
| Age Ranges | | Y | |
| Study Populations | | | Υ [1] |
| Concomitant Medications | | | |
| Concomitant Medications | | | Υ |

#### NOTES:

- Y = Yes display generated.
- 1. Listing includes only subjects excluded from any population.

#### 7. PRIMARY STATISTICAL ANALYSES

#### 7.1. Pharmacokinetic Analyses

#### 7.1.1. Overview of Planned Pharmacokinetic Analyses

The PK analyses will be based on the PK Population, unless otherwise specified.

Table 3 provides an overview of the planned analyses, with full details being presented in Appendix 10: List of Data Displays.

Table 3 Overview of Planned Pharmacokinetic Analyses

| Display Type | | Untransformed | | | | | | Ln-Transformed | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Stat | Stats Analysis | | Sumr | mmary Individual | | Stats Analysis | | ysis | Summary | | Individual | | |
| | Т | F | L | Т | F | F | L | Т | F | Г | Т | F | F | Г |
| PK Concentrations | | | | Υ | <b>Y</b> [1] [2] | <b>Y</b> [1] | Υ | | | | | | | |
| Plasma PK<br>Parameters | Υ | Υ | | Υ | <b>Y</b> [1] [2] | Υ | Υ | | | Υ | Υ | | | |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.
- [1] Linear and Semi-Logarithmic plots will be created on the same display.
- [2] Separate mean and median plots will be generated.

#### 7.1.2. Drug Concentration Measures

Refer to Appendix 3: Data Display Standards & Handling Conventions (Section 3 Reporting Process & Standards).

#### 7.1.3. Pharmacokinetic Parameters

#### 7.1.3.1. Deriving Pharmacokinetic Parameters

- Refer to Appendix 3: Data Display Standards & Handling Conventions (Section 3 Reporting Process & Standards).
- The PK parameters will be calculated by standard non-compartmental analysis according to current working practices and using Phoenix WinNonlin Version 6.4 or higher.
- All calculations of non-compartmental parameters will be based on actual sampling times.
- Pharmacokinetic parameters described in Table 4 will be determined from the plasma concentration-time data, as data permits.

Table 4 Derived Plasma Pharmacokinetic Parameters

| Parameter | Parameter Description |
|---|---|
| AUC(0-t) | Area under the concentration-time curve (AUC) from time 0 (predose) to time of the last quantifiable concentration, to be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| AUC0-24 | Area under the concentration-time curve (AUC) over time 0 (predose) to 24 hours after dose administration, to be calculated using the linear trapezoidal rule for each incremental trapezoid and the log trapezoidal rule for each decremental trapezoid. |
| AUC(0-∞) | Area under the concentration-time curve from time 0 (predose) extrapolated to infinite time, calculated as: $AUC(0-\infty) = AUC(0-t) + Ct / \lambda z$ |
| | where Ct is the last observed quantifiable concentration. |
| %AUCex | The percentage of AUC(0-∞) obtained by extrapolation (%AUCex) will be calculated as: |
| | [AUC(0-∞) – AUC(0-t)] / AUC(0-∞) x 100 |
| Cmax | Maximum observed concentration, determined directly from the concentration-time data. |
| Ct | The last observed quantifiable concentration |
| C24 | The observed concentration at 24 hours after dose administration |
| tmax | Time to first occurrence of Cmax |
| tlag | Lag time before observation of drug concentrations in sampled matrix |
| t½ | Terminal phase half-life will be calculated as: |
| | $t\frac{1}{2} = \ln 2 / \lambda z$ |
| λz | Terminal-phase rate constant |
| CL/F | The apparent oral clearance |
| Vz/F | The apparent volume of distribution during the terminal phase |

#### NOTES:

• Additional parameters may be included as required.

#### 7.1.3.2. Statistical Analysis of Pharmacokinetic Parameters

The following PK statistical analyses will only be performed, if sufficient data are available (i.e. if subjects have well defined plasma profiles).

# Pharmacokinetic Statistical Analyses Endpoint(s) Plasma primary PK endpoints include AUC(0-∞), AUC(0-t) and Cmax of DTG, as data permit Model Specification In Part 1 of this study, the In-transformed AUC(0-∞), AUC(0-t), and Cmax values for DTG will be analyzed separately using a mixed effects model, fitting fixed effect terms for period, and

#### **Pharmacokinetic Statistical Analyses**

treatment, and treating subject as a random effect. Point estimates and 90% CIs for the differences of interest (conventional DTG 5 x 10 mg tablets administered direct to mouth [Treatment A, Test] versus conventional DTG 1 x 50 mg tablet administered direct to mouth [Treatment B, Reference]) will be constructed using the residual variance

• In Part 2 of this study, the In-transformed AUC(0-∞), AUC(0-t), and Cmax values for DTG will be analyzed separately using a mixed effects model, fitting fixed effect terms for period and treatment, and treating subject as a random effect. Point estimates and 90% CIs for the differences of interest (5 x 5 mg dispersible DTG tablets [Treatment C, Test 1] versus conventional DTG 1 x 25 mg tablet administered direct to mouth [Treatment E, Reference], and conventional DTG 5 x 5 mg tablets administered direct to mouth [Treatment D, Test 2] versus conventional DTG 1 x 50 mg tablet administered direct to mouth [Treatment E, Reference]) will be constructed using the residual variance.

#### **Model Checking & Diagnostics**

Refer to Appendix 8: Model Checking and Diagnostics for Statistical Analyses.

#### **Model Results Presentation**

• Statistical analysis by ANOVA will be presented in tabular format with geometric mean ratios between TIVICAY™ conventional and dispersible tablets versus conventional DTG tablets, and 90% CIs for the ratios of AUC(0-∞), AUC(0-t) and Cmax for DTG.

Part 1 Example SAS Code:

PROC MIXED:

CLASS USUBJID TRTA APERIOD:

MODEL LOGPKPARM =TRTA APERIOD /DDFM=KR;

RANDOM USUBJID:

LSMEANS TRTA;

ESTIMATE 'A VS B' TRTA 1 -1/CL ALPHA=0.1;RUN;

Part 2 Example SAS Code:

PROC MIXED:

CLASS USUBJID TRTA APERIOD;

MODEL LOGPKPARM =TRTA APERIOD /DDFM=KR;

RANDOM USUBJID;

LSMEANS TRTA;

ESTIMATE 'C VS E' TRTA 1 0 -1/CL ALPHA=0.1;

ESTIMATE 'D VS E' TRTA 0 1 -1/CL ALPHA=0.1;RUN;

#### 7.1.4. Interim Analysis

#### 7.1.4.1. Overview of Planned Analyses

No interim analysis is planned for this study.

#### 8. SECONDARY STATISTICAL ANALYSES

#### 8.1. Safety Analyses

The safety analyses will be based on the "All Subjects" population, unless otherwise specified.

Table 5 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 10: List of Data Displays.

Table 5 Overview of Planned Safety Analyses

| Display Type | | Abso | olute | | Change from Baseline | | | |
|---|---|---|---|---|---|---|---|---|
| | Sum | ımary | Indiv | ridual | Sum | mary | Individual | |
| | T | F | F | L | T | F | F | L |
| Exposure | | | | | | | | |
| Exposure Data | | | | Υ | | | | |
| AEs | | | | | | | | |
| All AEs | Υ | | | Υ | | | | |
| All Drug-Related AEs | Υ | | | Υ | | | | |
| Common Non-serious AEs | Y | | | | | | | |
| Serious AEs | Υ | | | Υ | | | | |
| Withdrawal AEs | | | | Υ | | | | |
| Laboratory Values | | | | | | | | |
| Clinical Chemistry | | | | Υ [2] | Υ | | | |
| Hematology | | | | Y [2] | Υ | | | |
| Urinalysis (Dipstick) | Υ | | | Υ [2] | | | | |
| Electrocardiograms (E | CGs) | | | | | | | |
| ECG Findings | Υ | | | Υ [3] | | | | |
| ECG Values | | | | Υ [4] | | | | |
| Vital Signs | | | | | | | | |
| Vital Signs | | | | Y [4] | Υ | | | Y [4] |
| Liver | | | | | | | | |
| Liver Events [1] | | | | Υ | | | | |

#### NOTES:

- 1. Conditional display, it will only be produced when an event has occurred.
- 2. Displays contain only subjects with DAIDS toxicities for HIV-infected patients of Grade 2 or higher
- 3. Displays contain only subjects with abnormal findings
- 4. Displays contain only subjects with values of potential clinical importance
- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents TFL related to any displays of individual subject observed raw data.

#### 8.2. Exploratory Analyses

The exploratory analyses will be based on the "All Subjects" population, unless otherwise specified.

Table 6 provides an overview of the planned analyses, with further details of data displays being presented in Appendix 10: List of Data Displays.

Table 6 Overview of Planned Exploratory Analyses

| Display Type | Absolute | | | |
|---|---|---|---|---|
| | Sum | mary | Indiv | idual |
| | T | F | F | L |
| Palatability | | | | |
| Palatability Questionnaire Results | Y | | | Υ |

#### NOTES:

- T = Table, F = Figure, L = Listing, Y = Yes display generated.
- Stats Analysis = Represents TFL related to any formal statistical analyses (i.e. modelling) conducted.
- Summary = Represents TFL related to any summaries (i.e. descriptive statistics) of the observed raw data.
- Individual = Represents FL related to any displays of individual subject observed raw data.

#### 9. REFERENCES

GlaxoSmithKline Document Number 2016N302761\_00 (Original – 23-FEB-2017): A 2-Part Phase I, Single Dose, Crossover Relative Bioavailability Study of Both TIVICAY 10 mg Conventional Tablets and 5 mg Dispersible Tablets Compared to Conventional TIVICAY Tablets in Healthy Adult Subjects (23-FEB-2017)

# 10. APPENDICES

| Section | Appendix |
|---|---|
| RAP Section 5 | : General Considerations for Data Analyses & Data Handling Conventions |
| Section 10.1 | Appendix 1: Time and Events |
| Section 10.2 | Appendix 2: Treatment States & Phases |
| Section 10.3 | Appendix 3: Data Display Standards & Handling Conventions |
| | Study Treatment & Sub-group Display Descriptors |
| | Baseline Definitions & Derivations |
| | Reporting Process & Standards |
| Section 10.4 | Appendix 4: Derived and Transformed Data |
| | General, Study Population & Safety |
| | Pharmacokinetic |
| | Exploratory |
| Section 10.5 | Appendix 5: Premature Withdrawals & Handling of Missing Data |
| | Premature Withdrawals |
| | Handling of Missing Data |
| Section 10.6 | Appendix 6: Values of Potential Clinical Importance |
| Section 10.7 | Appendix 7: Multiple Comparisons and Multiplicity |
| Section 10.8 | Appendix 8: Model Checking and Diagnostics for Statistical Analyses |
| Other RAP App | endices |
| Section 10.9 | Appendix 9: Abbreviations & Trade Marks |
| Section 10.10 | Appendix 10: List of Data Displays |

# 10.1. Appendix 1: Time & Events

#### 10.1.1. Protocol Defined Time & Events

| | All Study Periods (Parts 1 and 2) | | | | | | dn | Notes Day -1 of Periods 2 -3 may be the same day as Day 6 of prior periods | |
|---|---|---|---|---|---|---|---|---|---|
| | | | Day | y 1 | Day 2 | Day 3 | Day 4 | Follow-up | At Follow-up – Male subjects with no ongoing AEs or |
| Assessments | Day -1 | Pre-dose | 0 hr | Post Dose | 24 hr | 48 hr | 72 hr | Fol | Vital Sign/Laboratory measures of clinical concern may be followed virtually by the site via telephone contact. |
| Admission to Unit | X | | | | | | | | |
| Discharge | | | | | | | Х | | |
| Outpatient Visit | | | | | | | | X | Follow-up visit will occur 7 to 10 days post last dose. |
| 12-lead ECG (single) | X | | | | | | | | |
| Vital signs | Х | Х | | | X | | Х | Х | Single vital sign measurements performed at all time points. |
| Brief Physical Exam | Х | | | | | | | | Drug/Alcohol/Cotinine/pregnancy will be performed per the |
| Urine Drug/Alcohol/Cotinine | Х | | | | | | ĺ | | standard practice of the site. |
| Pregnancy test (urine; WCBP) | Х | | | | | | | Х | <ul> <li>Clinical laboratory tests – see Protocol Table 5, Section 9.3.4.</li> <li>Clinical laboratory tests at follow-up are only necessary if</li> </ul> |
| Clinical laboratory tests | Х | | | | X | | | X* | subject had a previous abnormal lab value |
| Dosing | | | Χ | | | | į | | See Protocol Section 7.1 |
| Palatability Assessment | | | | Start w/in 10 min post-dose | | | | | Complete for each dispersion treatment C (see Protocol Section 12.8, Appendix 8) |
| PK Sampling | | Х | | Collect at: 0.5, 1, 1<br>24, 48 an | .5, 2, 2.5, 3<br>d 72 hrs po | s, 4, 5, 6, 8,<br>ost-dose. | 12, 16, | | Pre-dose (within 15 minutes prior to dosing), Protocol Section 9.4 |
| Meals | | from 10 hrs prior to Standard for the study center to 4 hrs post-dose | | | | tudy center | | | See also Protocol Section 6.3.2 and Section 6.3.3 |
| Adverse Events / SAE | X | ¢======== | | | | | | X | |
| Concomitant medications | X | <b>&lt;=====</b> | ←===========X======X=======< | | | | | | |

#### 10.2. Appendix 2: Treatment States and Phases

#### 10.2.1. Treatment States

Assessments and events will be classified according to time of occurrence relative to the start and/or stop date of the study treatment.

#### 10.2.1.1. Treatment States for Safety Data

| Treatment State | Definition |
|---|---|
| Pre-Treatment | Date/Time ≤ Study Treatment Start Date/Time |
| On-Treatment | Study Treatment Start Date/Time < Date/Time ≤ Study Treatment Stop Date/Time + 6 days |
| Post-Treatment | Date/Time > Study Treatment Stop Date/Time + 6 days |

#### NOTES:

• If the study treatment stop date is missing then the assessment will be considered to be On-Treatment

#### 10.2.1.2. Treatment States for AE Data

| Treatment State | Definition |
|---|---|
| Pre-Treatment | AE Start Date < Study Treatment Start Date |
| On-Treatment | If AE onset date is on or after treatment start date & on or before treatment stop date with 7 days lag time. |
| | Study Treatment Start Date ≤ AE Start Date ≤ Study Treatment Stop Date + 6 days |
| Post-Treatment | If AE onset date is after the treatment stop date with 6 days lag time. |
| | AE Start Date > Study Treatment Stop Date + 6 days |
| Onset Time | If Treatment Start Date > AE Onset Date = AE Onset Date – Treatment Start Date |
| Since 1st Dose | If Treatment Start Date ≤ AE Onset Date = AE Onset Date – Treatment Start Date +1 |
| (Days) | Missing otherwise. |
| Duration (Days) | AE Resolution Date – AE Onset Date + 1 |
| Drug-related | If relationship is marked 'YES' on eCRF OR value is missing. |

#### NOTES:

• If the study treatment stop date is missing then the AE will be considered to be On-Treatment.

# 10.3. Appendix 3: Data Display Standards & Handling Conventions

#### 10.3.1. Study Treatment & Sub-group Display Descriptors

| Treatment Group Descriptions | | | | |
|---|---|---|---|---|
| Study | | Treatment Group | Data Displays for Reporting | |
| Part | Code | Description | Description <sup>[1]</sup> | Order [2] |
| 1 | Α | DTG conventional 10 mg tablets (5 tablets) administered direct to mouth (test) | Treatment A | 1 |
| 1 | В | DTG conventional 50 mg tablet administered direct to mouth (reference) | Treatment B | 2 |
| 2 | С | DTG dispersible 5-mg tablets<br>(5 tablets) administered as a<br>dispersion and immediately taken<br>(test 1) | Treatment C | 3 |
| 2 | D | DTG dispersible 5-mg tablets (5 tablets) administered direct to mouth (test 2) | Treatment D | 4 |
| 2 | E | DTG conventional 25 mg tablet administered direct to mouth (reference) | Treatment E | 5 |

#### NOTES:

- 1. The word "Treatment" may be omitted from displays in order to limit wrapping
- 2. Order represents treatments being presented in TFL, as appropriate.

#### 10.3.2. Baseline Definition & Derivations

#### 10.3.2.1. Baseline Definitions

For all endpoints (except as noted in baseline definitions) the baseline value will be the latest pre-dose assessment. Baseline definitions are applicable to each period.

| Parameter | Study Assess | Study Assessments Considered As Baseline | | |
|---|---|---|---|---|
| | Screening | Day -1 | Day 1 (Pre-Dose) | Data Display |
| Safety | Safety | | | |
| Hematology | X | Χ | | Day -1 |
| Clinical Chemistry | X | Χ | | Day -1 |
| 12-Lead ECG | X | Χ | | Day -1 |
| Vital Signs | X | Χ | X | Day 1 (Pre-Dose) |

#### NOTES:

| Parameter | Study Assessments Considered As Baseline | | | Baseline Used in |
|---|---|---|---|---|
| | Screening | Day -1 | Day 1 (Pre-Dose) | Data Display |

 Unless otherwise stated, the mean of replicate assessments at any given time point will be used as the value for that time point.

#### 10.3.2.2. Derivations and Handling of Missing Baseline Data

| Definition | Reporting Details |
|----------------------|------------------------------------|
| Change from Baseline | = Post-Dose Visit Value – Baseline |

#### NOTES:

- Unless otherwise specified, the baseline definitions specified in Section 10.3.2.1 Baseline Definitions will be used for derivations for endpoints / parameters and indicated on summaries and listings.
- Unless otherwise stated, if baseline data is missing no derivation will be performed and will be set to missing.
- The baseline definition will be footnoted on all change from baseline displays.

#### 10.3.3. Reporting Process & Standards

#### **Reporting Process**

#### **Software**

The currently supported versions of SAS and Phoenix WinNonlin software will be used.

#### **Analysis Datasets**

- Analysis datasets will be created according to CDISC standards SDTM IG Version 3.1.3 & AdaM IG Version 1.0.
- For creation of AdaM datasets (ADCM/ADAE), the same version of dictionary datasets will be implemented for conversion from SI to SDTM.

#### **Generation of RTF Files**

RTF files will be generated for all reporting efforts described in the RAP.

#### **Reporting Standards**

#### General

- The current GSK IDSL will be applied for reporting, unless otherwise stated:
  - 4.03 to 4.23: General Principles
  - o 5.01 to 5.08: Principles Related to Data Listings
  - 6.01 to 6.11: Principles Related to Summary Tables
  - o 7.01 to 7.13: Principles Related to Graphics

#### **Formats**

- All data will be reported according to the actual treatment the subject received unless otherwise stated.
- GSK IDSL Statistical Principles (5.03 & 6.06.3) for decimal places will be adopted for reporting
  of data based on the raw data collected.
- Numeric data will be reported at the precision collected on the eCRF.
- The reported precision from non eCRF sources will follow the IDSL statistical principles but may be adjusted to a clinically interpretable number of DP's.

#### **Planned and Actual Time**

#### **Reporting Standards**

- Reporting for tables, figures and formal statistical analyses :
  - Planned time relative to dosing will be used in figures, summaries, statistical analyses and calculation of any derived parameters, unless otherwise stated.
  - The impact of any major deviation from the planned assessment times and/or scheduled visit days on the analyses and interpretation of the results will be assessed as appropriate.
- Reporting for Data Listings:
  - Planned and actual time relative to study drug dosing will be shown in listings (Refer to IDSL Statistical Principle 5.05.1).
  - Unscheduled or unplanned readings will be presented within the subject's listings.
  - Visits outside the protocol defined time-windows (i.e. recorded as protocol deviations) will be included in listings but omitted from figures, summaries and statistical analyses.

#### **Unscheduled Visits**

- Unscheduled visits will not be included in summary tables.
- Unscheduled visits will not be included in figures.
- All unscheduled visits will be included in listings.

**Reporting of Pharmacokinetic Parameters** 

#### **Descriptive Summary Statistics** Continuous Data Refer to IDSL Statistical Principle 6.06.1 NQs at the beginning of a subject profile (i.e. before the first incidence of a measurable concentration) are deemed to be zero as it is assumed that in this circumstance no drug is yet measurable in the blood. For NQs at the end of the subject profile (i.e. after the last incidence of a measurable concentration); for individual plots and pharmacokinetic analyses these are dropped (set to missing) as they do not provide any useful information (and can erroneously indicate that absolutely no drug is present) for summary statistics these are set to 0 (to avoid skewing of the summary statistics) Individual NQs which fall between two measurable concentrations are set to missing (individual values of this nature are assumed to be an anomaly) If two or more NQ values occur in succession between measurable concentrations, the profile will be deemed to have terminated at the last measurable concentration prior to these NQs. For the purpose of individual subject plots, these NQs will be set to 0, and the subsequent measurable concentrations will be retained. For the derivation of pharmacokinetic parameters, these NQs and any subsequent measurable concentrations will be omitted (set to missing). Categorical Data N (number of subjects in subgroup), n (number of subjects with evaluable data), frequency, % Reporting of Pharmacokinetic Concentration Data Descriptive Refer to IDSL Statistical Principle 6.06.1 **Summary Statistics** Assign zero to NQ values (Refer to GUI\_51487 for further details)

| Reporting Standards | |
|---|---|
| Descriptive<br>Summary Statistics<br>(Ln-Transformed) | N (number of subjects in subgroup), n (number of subjects with evaluable data), geometric mean, 95% CI of geometric mean, standard deviation (SD) of logged data and between geometric coefficient of variation (CVb (%)) will be reported. $ \text{CV}_b \text{ (\%)} = \sqrt{\left(\text{exp}(\text{SD}^2) - 1\right) * 100} \\ \text{(SD = SD of In-transformed data)} $ |
| Parameters Not<br>Being Ln-<br>Transformed | tmax, tlag, first point, last point, and number of points used in the determination of $\lambda z$ , %AUCex. |
| Summary Tables The following PK parameters will not be summarised: first point, last point, and number of points used in the determination of λz | |
| Listings | Include the first point, last point and number of points used in the determination of $\lambda z$ . |
| Graphical Displays | |
| Refer to IDSL Statistical Principals 7.01 to 7.13. | |

#### 10.4. Appendix 4: Derived and Transformed Data

#### 10.4.1. General

#### **Multiple Measurements at One Time Point**

- Mean of the measurements will be calculated and used in any derivation of summary statistics but if listed, all data will be presented.
- If there are two values within a time window the value closest to the target day for that window will be used. If values are the same distance from the target then the mean will be taken.
- Subjects having both High and Low values for Normal Ranges at any post-baseline visits for safety parameters will be counted in both the High and Low categories of "Any visit postbaseline" row of related summary tables. This will also be applicable to relevant Potential Clinical Importance summary tables.

#### Study Day

- Calculated as the number of days from randomisation date :
  - Ref Date = Missing → Study Day = Missing
  - Ref Date < Randomisation Date → Study Day = Ref Date Randomisation Date</li>
  - Ref Data ≥ Randomisation Date → Study Day = Ref Date (Randomisation Date) + 1

#### 10.4.2. Study Population

#### **Demographics**

#### Age

- GSK standard IDSL algorithms will be used for calculating age where birth date will be imputed as follows:
  - Only the year of birth will be collected. The date and month will be imputed as '30th June'.
- Birth date will be presented in listings as 'YYYY'.

#### **Body Mass Index (BMI)**

Calculated as Weight (kg) / [Height (m)<sup>2</sup>]

#### 10.4.3. Safety

#### **ECG Parameters**

#### RR Interval

- IF RR interval (msec) is not provided directly, then RR can be derived as :
  - [1] If QTcB is machine read & QTcF is not provided, then:

$$RR = \left[ \left( \frac{QT}{QTcB} \right)^2 \right] * 1000$$

[2] If QTcF is machine read and QTcB is not provided, then:

$$RR = \left[ \left( \frac{QT}{QT cF} \right)^2 \right] * 1000$$

 If ECGs are manually read, the RR value preceding the measurement QT interval should be a collected value THEN do not derive.

#### **ECG Parameters**

• Machine read values of RR should not be replaced with derived values.

#### **Corrected QT Intervals**

- When not entered directly in the eCRF, corrected QT intervals by Bazett's (QTcB) and Fredericia's (QTcF) formulas will be calculated, in msec, depending on the availability of other measurements.
- IF RR interval (msec) is provided then missing QTcB and/or QTcF will be derived as :

$$QTcB = \frac{QT}{\sqrt{\frac{RR}{1000}}}$$

$$QTcF = \frac{QT}{3\sqrt{\frac{RR}{1000}}}$$

#### AEs

#### **AEs OF Special Interest**

- Hypersensitivity reaction (HSR) and rash
- Liver Events
- Renal Function
- Creatine Phosphokinase (CPK) elevations

# 10.5. Appendix 5: Premature Withdrawals & Handling of Missing Data

#### 10.5.1. Premature Withdrawals

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Subject study completion (i.e. as specified in the protocol) was defined as completing all phases of the study including the follow-up visit.</li> <li>Withdrawn subjects may be replaced in the study.</li> <li>All available data from subjects who were withdrawn from the study will be listed and all available planned data will be included in summary tables and figures, unless otherwise specified.</li> </ul> |

# 10.5.2. Handling of Missing Data

| Element | Reporting Detail |
|---|---|
| General | <ul> <li>Missing data occurs when any requested data is not provided, leading to blank fields on the collection instrument:</li> <li>These data will be indicated by the use of a "blank" in subject listing displays. Unless all data for a specific visit are missing in which case the data is excluded from the table.</li> </ul> |
| | <ul> <li>Answers such as "Not applicable" and "Not evaluable" are not considered to<br/>be missing data and should be displayed as such.</li> </ul> |
| Outliers | Any subjects excluded from the summaries and/or statistical analyses will be documented along with the reason for exclusion in the clinical study report. |

#### 10.5.2.1. Handling of Missing Dates

| Element | Reporting Detail |
|---|---|
| General | Partial dates will be displayed as captured in subject listing displays. |
| AEs | <ul> <li>The eCRF allows for the possibility of partial dates (i.e., only month and year) to be recorded for AE start and end dates; that is, the day of the month may be missing. In such a case, the following conventions will be applied for calculating the time to onset and the duration of the event: <ul> <li>Missing Start Day: First of the month will be used unless this is before the start date of study treatment; in this case the study treatment start date will be used and hence the event is considered On-treatment as per Appendix 2: Treatment States and Phases.</li> <li>Missing Stop Day: Last day of the month will be used, unless this is after the stop date of study treatment; in this case the study treatment stop date will be used.</li> </ul> </li> <li>Completely missing start or end dates will remain missing, with no imputation applied. Consequently, time to onset and duration of such events will be missing.</li> </ul> |

| Element | Reporting Detail |
|---|---|
| | Start or end dates which are completely missing (i.e. no year specified) will |
| | remain missing, with no imputation applied. |

# 10.5.2.2. Handling of Partial Dates

| Element | Reporting Detail |
|---|---|
| Concomitant<br>Medications | <ul> <li>Partial dates for any concomitant medications recorded in the eCRF will be imputed using the following convention:</li> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> <li>The recorded partial date will be displayed in listings.</li> </ul> |
| AEs | <ul> <li>Any partial dates for AEs will be raised to data management. If the full date cannot be ascertained, the following assumptions will be made: <ul> <li>If the partial date is a start date, a '01' will be used for the day and 'Jan' will be used for the month.</li> <li>However, if these results in a date prior to Week 1 Day 1 and the event could possibly have occurred during treatment from the partial information, then the Week 1 Day 1 date will be assumed to be the start date.</li> <li>The AE will then be considered to start on-treatment (worst case).</li> <li>If the partial date is a stop date, a '28/29/30/31' will be used for the day (dependent on the month and year) and 'Dec' will be used for the month.</li> </ul> </li> <li>The recorded partial date will be displayed in listings.</li> </ul> |

| Element | Reporting Detail |
|---------|-----------------------------------------------------|
| 10.6. | Appendix 6: Values of Potential Clinical Importance |

#### 10.6.1. **ECG**

| ECG Parameter Units | | Potential Clinically Important Range | |
|---|---|---|---|
| | | Lower | Upper |
| Absolute | | | |
| | | > 450[1] | |
| Abaqluta OTa Interval | | > 450[2] | ≤ 479 <sup>[2]</sup> |
| Absolute QTc Interval | msec | ≥ 480[2] | ≤ 499 <sup>[2]</sup> |
| | | ≥ 500 <sup>[2]</sup> | |
| Absolute PR Interval | msec | < 110[1] | > 220[1] |
| Absolute QRS Interval | msec | < 75 <sup>[1]</sup> | > 110 <sup>[1]</sup> |
| Change from Baseline | | | |
| | msec | ≤ 30 <sup>[2]</sup> | |
| Increase from Baseline QTc | msec | > 30[2] | ≤ 59 <sup>[2]</sup> |
| | msec | ≥ 60[1] | |

#### NOTES:

- Represent standard ECG values of PCI for HV studies.
   Represent further subdivisions of ECG values for analysis.

#### 10.6.2. **Vital Signs**

| Vital Sign Parameter | Units | Potential Clinically | Important Range |
|--------------------------|-------|----------------------|-----------------|
| (Absolute) | | Lower | Upper |
| Systolic Blood Pressure | mmHg | < 85 | > 160 |
| Diastolic Blood Pressure | mmHg | < 45 | > 100 |
| Heart Rate | bpm | < 40 | > 110 |

# 10.7. Appendix 7: Multiple Comparisons & Multiplicity

# 10.7.1. Handling of Multiple Comparisons & Multiplicity

No adjustments for multiplicity will be made.

# 10.8. Appendix 8: Model Checking and Diagnostics for Statistical Analyses

#### 10.8.1. Statistical Analysis Assumptions

| Endpoint(s) | <ul> <li>PK endpoints AUC(0-∞), AUC(0-t) and Cmax</li> </ul> |
|-------------|--------------------------------------------------------------|
| Analysis | Mixed Effects |

#### **Assumptions:**

- Model assumptions will be applied, but appropriate adjustments may be made based on the data
- The Kenward and Roger method for approximating the denominator degrees of freedom and correcting for bias in the estimated variance-covariance of the fixed effects will be used.

# 10.9. Appendix 9 – Abbreviations & Trade Marks

#### 10.9.1. Abbreviations

| Abbreviation | Description |
|---|---|
| ADaM | Analysis Data Model |
| AE | Adverse Event |
| AUC(0-t) | Area under the concentration-time curve (AUC) from time 0 (predose) |
| | to time of the last quantifiable concentration |
| AUC0-24 | Area under the concentration-time curve (AUC) over time 0 (predose) |
| | to 24 hours after dose administration |
| $AUC(0-\infty)$ | Area under the concentration-time curve from time 0 (predose) |
| | extrapolated to infinite time |
| %AUCex | The percentage of AUC( $0-\infty$ ) obtained by extrapolation |
| BA | Bioavailability |
| BMI | Body Mass Index |
| C24 | The observed concentration at 24 hours after dose administration |
| CDISC | Clinical Data Interchange Standards Consortium |
| CL/F | The apparent oral clearance |
| Cmax | Maximum observed concentration |
| CI | Confidence Interval |
| CPK | Creatine Phosphokinase |
| Ct | The last observed quantifiable concentration |
| CVb | Coefficient of Variation (Between) |
| DAIDS | Division of Acquired Immune Deficiency Syndrome |
| DTG | Dolutegravir |
| ECG | Electrocardiogram |
| eCRF | Electronic Case Report Form |
| GSK | GlaxoSmithKline |
| HSR | Hypersensitivity reaction |
| ICH | International Conference on Harmonisation |
| IDSL | Integrated Data Standards Library |
| kg | Kilograms |
| m | Meters |
| mg | Milligrams |
| msec | Milliseconds |
| PK | Pharmacokinetic |
| QTcF | Fridericia's QT Interval Corrected for Heart Rate |
| QTcB | Bazett's QT Interval Corrected for Heart Rate |
| R&D | Research and Development |
| RAP | Reporting & Analysis Plan |
| SAC | Statistical Analysis Complete |
| SAS | Statistical Analysis Software |
| SD | Standard deviation |
| SDTM | Study Data Tabulation Model |
| TFL | Tables, Figures & Listings |

| Abbreviation | Description |
|---|---|
| t½ | Terminal phase half-life |
| tlag | Lag time before observation of drug concentrations in sampled matrix |
| tmax | Time to first occurrence of Cmax |
| Vz/F | The apparent volume of distribution during the terminal phase |
| λz | Terminal-phase rate constant |

#### 10.9.2. Trademarks

| Trademarks of the GlaxoSmithKline<br>Group of Companies |
|---------------------------------------------------------|
| TIVICAY |

| Trademarks not owned by the GlaxoSmithKline Group of Companies |
|----------------------------------------------------------------|
| Phoenix WinNonlin |
| SAS |

#### 10.10. Appendix 10: List of Data Displays

The following numbering will be applied for RAP generated displays:

| Section | Tables | Figures |
|----------------------------|------------|------------|
| Study Population | 1.1 to 1.8 | NA |
| Safety | 2.1 to 2.9 | NA |
| Pharmacokinetic | 3.1 to 3.5 | 3.1 to 3.7 |
| Exploratory (Palatability) | 4.1 | NA |
| Section Listings | | ings |
| ICH Listings | 1 to 38 | |

#### 10.10.1. Mock Example Shell Referencing

Non IDSL specifications will be referenced as indicated.

| Section | Figure | Table | Listing |
|----------------------------|---------|---------|---------|
| Study Population | POP_Fn | POP_Tn | POP_Ln |
| Safety | SAFE_Fn | SAFE_Tn | SAFE_Ln |
| Pharmacokinetic | PK_Fn | PK_Tn | PK_Ln |
| Exploratory (Palatability) | EXP_Fn | EXP_Tn | EXP_Ln |

#### NOTES:

Non-Standard displays are indicated in the 'IDSL / TST ID / Example Shell' or 'Programming Notes' column as '[Non-Standard] + Reference.'

#### 10.10.2. Deliverable [Priority]

| Delivery [Priority] [1] | Description |
|-------------------------|-------------------------------------|
| SAC [X] | Final Statistical Analysis Complete |

#### NOTES:

1. Indicates priority (i.e. order) in which displays will be generated for the reporting effort.

# 10.10.3. Study Population Tables

| Study F | Study Population Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Subject | Disposition ar | nd Analysis Sets | | | |
| 1.1 | All Subjects | NS1 | Summary of Number of Subjects Enrolled by Country and Site ID | | SAC [1] |
| 1.2 | All Subjects | ES1 | Summary of Subject Disposition | | SAC [1] |
| 1.3 | Screened | ES6 | Summary of Reasons for Screening Failures | | SAC [1] |
| 1.4 | Screened | DV1 | Summary of Important Protocol Deviations | | SAC [1] |
| Demog | raphics | | | | |
| 1.5 | All Subjects | DM1 | Summary of Demographic Characteristics | | SAC [1] |
| 1.6 | All Subjects | DM5 | Summary of Race and Racial Combinations | | SAC [1] |
| 1.7 | All Subjects | DM6 | Summary of Race and Racial Combinations Details | | SAC [1] |
| 1.8 | All Subjects | DM11 | Summary of Age Ranges | | SAC[1] |

# 10.10.4. Safety Tables

| Safety | : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| AEs | | | | | |
| 2.1 | All Subjects | AE1 | Summary of All Adverse Events | | SAC [1] |
| 2.2 | All Subjects | AE1 | Summary of All Drug-Related Adverse Events | | SAC [1] |
| 2.3 | All Subjects | AE15 | Summary of Common (>=5%) Non-serious Adverse Events by System Organ Class and Preferred Term | | SAC [1] |
| 2.4 | All Subjects | AE16 | Summary of Serious Adverse Events by System Organ Class and Preferred Term | | SAC[1] |
| Labora | tory Values | | | | • |
| 2.5 | All Subjects | LB1 | Summary of Clinical Chemistry Values Change from Baseline | | SAC [1] |
| 2.6 | All Subjects | LB1 | Summary of Haematology Values Change from Baseline | | SAC [1] |
| 2.7 | All Subjects | UR3 | Summary of Urinalysis Dipstick Results | | SAC [1] |
| Electro | cardiograms | | | | |
| 2.8 | All Subjects | EG1 | Summary of ECG Findings | | SAC [1] |
| Vital Si | gns | | | | |
| 2.9 | All Subjects | VS1 | Summary of Change from Baseline in Vital Signs | | SAC[1] |

# 10.10.5. Pharmacokinetic Tables

| Pharma | acokinetic : Tal | oles | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| PK Co | ncentration Dat | a | | | |
| 3.1 | PK | PKCT1 | Summary of DTG Plasma Pharmacokinetic Concentration-Time Data by Study Part and Treatment | | SAC [1] |
| PK Der | ived Parameter | rs | | , | - |
| 3.2 | PK | PKPT4 | Summary of Derived DTG Plasma Pharmacokinetic Parameters (Non-Transformed) by Study Part and Treatment | Parameters with units | SAC [1] |
| 3.3 | PK | PKPT4 | Summary of Derived DTG Plasma Pharmacokinetic Parameters (Ln-Transformed) by Study Part and Treatment | Parameters with units | SAC [1] |
| PK Ana | alysis Tables | | | , | - |
| 3.4 | PK | PKPT3 | Statistical Analysis of DTG Plasma Pharmacokinetic Parameters, Study Part 1 | AUC(0-t), AUC(0-∞), and Cmax only by Treatment. Part 1 only. | SAC [1] |
| 3.5 | PK | PKPT3 | Statistical Analysis of DTG Plasma Pharmacokinetic Parameters, Study Part 2 | AUC(0-t), AUC(0-∞), and Cmax only by Treatment. Part 2 only. | SAC [1] |

# 10.10.6. Pharmacokinetic Figures

| Pharma | Pharmacokinetic : Figures | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Individ | ual Concentrati | on Plots | | | |
| 3.1 | PK | PKCF1X | Individual DTG Plasma Concentration-Time Plots by Subject (Linear and Semi-Logarithmic) | Paginate by Subject | SAC [1] |
| Mean / | Median Concer | ntration Plots | | | |
| 3.2 | PK | PKCF2 | Mean DTG Plasma Concentration-Time Plots by Treatment (Linear and Semi-Logarithmic) | All treatments for each Part on one page | SAC [1] |
| 3.3 | PK | PKCF3 | Median DTG Plasma Concentration-Time Plots by Treatment (Linear and Semi-Logarithmic) | All treatments for each Part on one page | SAC [1] |
| PK Ana | lysis Plots | | | | |
| 3.4 | PK | PKPF3 | Comparative Plot of Individual DTG Plasma Cmax by Treatment (Linear and Semi-Logarithmic) | All treatments for each Part on one page | SAC [1] |
| 3.5 | PK | PKPF3 | Comparative Plot of Individual DTG Plasma AUC(0-t) by Treatment (Linear and Semi-Logarithmic) | All treatments for each Part on one page | SAC [1] |
| 3.6 | PK | PKPF3 | Comparative Plot of Individual DTG Plasma AUC(0-∞) by Treatment (Linear and Semi-Logarithmic) | All treatments for each Part on one page | SAC [1] |
| 3.7 | PK | PKPF3 | Comparative Plot of Individual DTG Plasma C24 by Treatment (Linear and Semi-Logarithmic) | All treatments for each Part on one page | SAC [1] |

# 10.10.7. Exploratory Tables

| Explora | Exploratory : Tables | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Palatab | Palatability | | | | |
| 4.1 | All Subjects | EXP_T1 | Summary of Palatability Questionnaire Results (Part 2, Treatment C Only) | | SAC[1] |

# 10.10.8. ICH Listings

| ICH : Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Rando | misation | | | • | |
| 1 | All Subjects | CP_TA1 | Listing of Randomised and Actual Treatment | | SAC [1] |
| Subjec | t Disposition | | | | |
| 2 | All Subjects | ES2 | Listing of Reasons for Study Withdrawal | | SAC [1] |
| 3 | Screened | ES7 | Listing of Reasons for Screening Failure | | SAC [1] |
| 4 | Screened | DV2 | Listing of Important Protocol Deviations | | SAC [1] |
| 5 | All Subjects | IE4 | Listing of Subjects with Inclusion/Exclusion Criteria Deviations | | SAC[1] |
| 6 | Screened | SP3 | Listing of Subjects Excluded from Any Population | | SAC [1] |
| Demographics | | | | | |
| 7 | All Subjects | DM4 | Listing of Demographic Characteristics | | SAC [1] |
| 8 | All Subjects | DM10 | Listing of Race | | SAC [1] |

| ICH : Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Conco | mitant Medicati | ons | | | |
| 9 | All Subjects | CM4 | Listing of Concomitant Medications | | SAC[1] |
| Exposi | ure | | | | |
| 10 | All Subjects | SAFE_L1 | Listing of Exposure Data | | SAC[1] |
| AEs | | | | | |
| 11 | All Subjects | AE2 | Listing of Relationship Between System Organ Class and Verbatim Text | | SAC[1] |
| 12 | All Subjects | AE7 | Listing of Subject Numbers for Individual Adverse Events | | SAC[1] |
| 13 | All Subjects | AE9CP | Listing of All Adverse Events | | SAC[1] |
| 14 | All Subjects | AE9CP | Listing of Study Drug Related Adverse Events | | SAC[1] |
| 15 | All Subjects | SAFE_L2 | Listing of Serious Adverse Events | | SAC[1] |
| 16 | All Subjects | AE9CP | Listing of Adverse Events Leading to Withdrawal from Study Drug | | SAC[1] |
| 17 | All Subjects | SAFE_L3 | Listing of Liver Adverse Events | | SAC[1] |

| ICH : Listings | | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Labora | tory Values | | | | |
| 18 | All Subjects | LB6 | Listing of Clinical Chemistry Toxicities of Grade 2 or Higher | | SAC [1] |
| 19 | All Subjects | LB6 | Listing of All Clinical Chemistry Data for Subjects with Toxicities of Grade 2 or Higher | | SAC [1] |
| 20 | All Subjects | LB6 | Listing of Haematology Toxicities of Grade 2 or Higher | | SAC [1] |
| 21 | All Subjects | LB6 | Listing of All Haematology Data for Subjects with Toxicities of Grade 2 or Higher | | SAC [1] |
| 22 | All Subjects | LB6 | Listing of Urinalysis Toxicities of Grade 2 or Higher | | SAC [1] |
| 23 | All Subjects | LB6 | Listing of All Urinalysis Data for Subjects with Toxicities of Grade 2 or Higher | | SAC [1] |
| Electro | cardiograms | | | | |
| 24 | All Subjects | EG6 | Listing of Abnormal ECG Findings | | SAC [1] |
| 25 | All Subjects | EG6 | Listing of All ECG Findings for Subjects with an Abnormal Finding | | SAC [1] |
| 26 | All Subjects | EG4 | Listing of ECG Values of Potential Clinical Importance | | SAC [1] |
| 27 | All Subjects | EG4 | Listing of All ECG Values for Subjects with Any Value of Potential Clinical Importance | | SAC[1] |

| ICH : L | ICH : Listings | | | | |
|---|---|---|---|---|---|
| No. | Population | IDSL / TST ID /<br>Example Shell | Title | Programming Notes | Deliverable<br>[Priority] |
| Vital Si | gns | | | | |
| 28 | All Subjects | VS5 | Listing of Vital Signs of Potential Clinical Importance | | SAC [1] |
| 29 | All Subjects | VS5 | Listing of All Vital Signs for Subjects with Potential Clinical Importance Values | | SAC [1] |
| Liver E | vent | | | | |
| 30 | All Subjects | LIVER5 | Listing of Liver Monitoring/Stopping Event Reporting | | SAC[1] |
| 31 | All Subjects | MH3 | Listing of Medical Conditions for Subjects with Liver Stopping<br>Events | | SAC[1] |
| 32 | All Subjects | SAFE_L5 | Listing of Alcohol Intake at Onset of Liver Event | | SAC[1] |
| 33 | All Subjects | PKCL1X | Listing of Plasma Concentration Data for Subjects with Liver Stopping Events | | SAC[1] |
| 34 | All Subjects | LIVER7 | Listing of Liver Biopsy Details | | SAC[1] |
| 35 | All Subjects | LIVER8 | Listing of Liver Imaging Details | | SAC[1] |
| Pharma | acokinetic | | | | |
| 36 | PK | PKCL1X | Listing of DTG Plasma Pharmacokinetic Concentration-Time Data by Treatment | Please list all the concentration data including unscheduled. Repeat for all treatments and Parts. | SAC [1] |
| 37 | PK | PKPL1X | Listing of Derived DTG Plasma Pharmacokinetic Parameters by Treatment | Repeat for all treatments and Parts. | SAC [1] |
| Explora | atory | | | | |
| 38 | All Subjects | EXP_L1 | Listing of Palatability Questionnaire Results (Part 2, Treatment C Only) | | SAC[1] |